CLINICAL TRIAL: NCT01083043
Title: Glycemic Variability Predicts Endothelial Dysfunction
Brief Title: Continuous Glucose Monitoring in Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 06035
Record Dates: First submitted 2010-03-05; First posted 2010-03-09 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Vascular Complications
Keywords: Glycemic Variability; Endothelial Dysfunction
MeSH Terms: conditions — Diabetic Angiopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus

SUMMARY:
It is well known that lowering average blood glucose decreases the risk of diabetic complications involving the small vessels, such as those found in the eyes, nerves and kidney. It is less clear however, if controlling fluctuations in blood glucose will further help to prevent such complications.

The purpose of this study is to examine the relationship between extreme fluctuations in glucose and damage to the blood vessel lining.

DETAILED DESCRIPTION:
Studies have shown that glycemic variability is associated with oxidative stress which in turn has been correlated with endothelial damage. Further, endothelial damage has been identified as a critical event lending way to the vascular complications seen in many disease states.

The specific aim of this study is to investigate the relationship between short-term glycemic variability and biomarkers of endothelial dysfunction while analyzing the influence of different variables and adjusting for covariates.

Data obtained from a continuous glucose monitoring system(CGMS), a device that continuously records interstitial glucose for a 72 hour period, is used to calculate glycemic variability. Serology for the determination of endothelial dysfunction biomarkers is obtained on day three.

Pearson and Spearman Rank Order correlations are utilized to determine whether there are any significant correlations between measures of glycemic variability and biomarker levels of endothelial dysfunction. Multiple regression analysis would also determine if glycemic variability predicts elevated biomarker levels even after controlling for other variables.

Provided the high prevalence of diabetic complications and their staggering socioeconomic costs, it is important to elucidate the relationship between glycemic variability and endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with Type 2 Diabetes Mellitus and glycosylated hemoglobin <8.0%

Exclusion Criteria:

* Age <18 or >65
* BMI >35
* Pregnant
* Baseline glycosylated hemoglobin <6.0% or >8.0%
* Winthrop University Hospital Employee or Staff member
* Vulnerable subject
* Uncontrolled hypertension(defined as systolic blood pressure >130 or diastolic blood pressure >80mmHg)
* Uncontrolled dyslipidemia (defined as LDL >130mg/dL; HDL <30mg/dL or triglycerides >199mg/dL)
* Current smoker or significant smoke exposure(defined as greater than 2 hours of exposure to second-hand smoke within the preceding 48hrs)
* Sympathomimetic use within the past week
* History of cardiovascular disease
* History of paroxysmal nocturnal hemoglobinuria
* History of thrombotic thrombocytopenic purpura
* History of stage II-V Chronic Kidney Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects with Type 2 Diabetes Mellitus from an outpatient Endocrinology Practice
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2006-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Serum levels of endothelial dysfunction biomarkers and glycemic variability | Day 3 of study enrollment
  The following biomarkers are studied: soluble e-selectin, vascular cell adhesion molecule-1, intercellular adhesion molecule-1 and asymmetric dimethylarginine. These analytes are highly correlated to endothelial dysfunction.

SECONDARY OUTCOMES:
Metabolic parameters and glycemic variability | Day 3 of study enrollment
  Blood pressure, body mass index, fasting glucose, highly sensitive CRP, HbA1c, lipid panel, adiponectin level, urine microalbumin/creatinine ratio will be measured and correlated to glycemic variability.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence E Shapiro, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Brownlee M. The pathobiology of diabetic complications: a unifying mechanism. Diabetes. 2005 Jun;54(6):1615-25. doi: 10.2337/diabetes.54.6.1615. No abstract available. PMID 15919781
- [Background] Lopes-Virella MF, Carter RE, Gilbert GE, Klein RL, Jaffa M, Jenkins AJ, Lyons TJ, Garvey WT, Virella G; Diabetes Control and Complications Trial/Epidemiology of Diabetes Intervention and Complications Cohort Study Group. Risk factors related to inflammation and endothelial dysfunction in the DCCT/EDIC cohort and their relationship with nephropathy and macrovascular complications. Diabetes Care. 2008 Oct;31(10):2006-12. doi: 10.2337/dc08-0659. Epub 2008 Jul 15. PMID 18628568
- [Background] Albertini JP, Valensi P, Lormeau B, Aurousseau MH, Ferriere F, Attali JR, Gattegno L. Elevated concentrations of soluble E-selectin and vascular cell adhesion molecule-1 in NIDDM. Effect of intensive insulin treatment. Diabetes Care. 1998 Jun;21(6):1008-13. doi: 10.2337/diacare.21.6.1008. PMID 9614623
- [Background] Krzyzanowska K, Mittermayer F, Wolzt M, Schernthaner G. Asymmetric dimethylarginine predicts cardiovascular events in patients with type 2 diabetes. Diabetes Care. 2007 Jul;30(7):1834-9. doi: 10.2337/dc07-0019. Epub 2007 Apr 24. PMID 17456842
- [Background] Schram MT, Chaturvedi N, Schalkwijk C, Giorgino F, Ebeling P, Fuller JH, Stehouwer CD; EURODIAB Prospective Complications Study. Vascular risk factors and markers of endothelial function as determinants of inflammatory markers in type 1 diabetes: the EURODIAB Prospective Complications Study. Diabetes Care. 2003 Jul;26(7):2165-73. doi: 10.2337/diacare.26.7.2165. PMID 12832330
- [Background] Meigs JB, Hu FB, Rifai N, Manson JE. Biomarkers of endothelial dysfunction and risk of type 2 diabetes mellitus. JAMA. 2004 Apr 28;291(16):1978-86. doi: 10.1001/jama.291.16.1978. PMID 15113816